CLINICAL TRIAL: NCT06544070
Title: Capillary Blood Accuracy
Acronym: CAPYBARA
Status: Not yet recruiting | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CTM-PRO-00028; 347665 (Other: IRAS ID)
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1: Participants who have undergone a laboratory FBC test that has returned a neutrophil count of ≤ 1.0 x109/L who can be consented within 24 hours of the result.
  Participants will donate one finger prick sample up to once per day to be tested on the Liberty device.
  Interventions: Device: Entia Liberty System
- Phase 2: Participants who have undergone a laboratory FBC test that has returned a neutrophil count of ≤ 1.5 x109/L who can be consented within 24 hours of the result.
  Participants will donate up to 3 finger prick samples to be tested on the Liberty device in a single session.
  Interventions: Device: Entia Liberty System
- Phase 3: Participants who are undergoing a routine venous draw as part of the standard of care as part of SACT toxicity monitoring.
  Participants will donate up to 3 finger prick samples to be tested on the Liberty device in a single session.
  Interventions: Device: Entia Liberty System

INTERVENTIONS:
Device: Entia Liberty System — Participants will donate finger-prick blood samples to be tested on the Entia Liberty System. The results will not be used to inform clinical decisions or affect routine clinical care in any way.

SUMMARY:
Entia is a health technology company that has developed a blood testing device called Entia Liberty, which analyses blood collected by a finger prick. Entia is sponsoring this research study to compare the results from Entia Liberty finger prick tests to results from the gold-standard laboratory analyser that tests blood from the arm, port, or PICC line.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of study entry
* Patients undergoing systemic anti-cancer therapy (SACT)
* Patients capable of providing written informed consent
* Patients undergoing routine Full Blood Count (FBC) laboratory blood tests as part of the standard of care

Additional inclusion criteria:

* Phase 1 (Longitudinal, low count data): Neutrophil Count ≤ 1.0 x109/L within 24 hours preceding consenting
* Phase 2 (Low count data): Neutrophil Count ≤ 1.5 x109/L within 24 hours preceding consenting

Exclusion Criteria:

* History or current diagnosis of haematological malignancy
* Inadequate use and understanding of the English language, requiring a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of solid tumour cancer who are undergoing systemic anti-cancer therapy (SACT).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Validity of of the Liberty System for haematological parameters of interest: Hb, WBC, PLT, ANC | Through study completion, up to 8 days per participant.
  The accuracy of the Liberty System will be measured by comparing the results of finger-prick blood samples that have been analysed using the Liberty System to the results of venous (blood from the arm, port or PICC line) blood samples that have been analysed by a standard laboratory haematology analyser.
Reliability of of the Liberty System for haematological parameters of interest: Hb, WBC, PLT, ANC | Through study completion, up to 8 days per participant.
  To measure the precision of the Liberty System by comparing the results of finger-prick blood samples that have been analysed by the Liberty System to each other, and to venous (blood from the arm, port or PICC line) blood samples that have been analysed by the Liberty System.

IPD SHARING:
Plan to Share IPD: No